CLINICAL TRIAL: NCT03788135
Title: Effect of Localized Muscle Cooling on Balance in Healthy Individuals
Brief Title: Localized Muscle Cooling on Balance in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Shahnawaz Anwer, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RRC-2018-011
Record Dates: First submitted 2018-12-20; First posted 2018-12-27 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Healthy
MeSH Terms: interventions — Cool-Down Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Quadriceps cooling (Experimental): Participants in this group will receive a cold pack on anterior thigh muscles for 20 minutes.
  Interventions: Behavioral: cooling
- Hamstring cooling (Experimental): Participants in this group will receive a cold pack on posterior thigh muscles for 20 minutes.
  Interventions: Behavioral: cooling
- Calf cooling (Experimental): Participants in this group will receive a cold pack on posterior leg muscles for 20 minutes.
  Interventions: Behavioral: cooling
- Back cooling (Experimental): Participants in this group will receive a cold pack on posterior low back muscles for 20 minutes.
  Interventions: Behavioral: cooling
- Control (No Intervention): The participants in the control group will be rested for 20 minutes without any intervention.

INTERVENTIONS:
Behavioral: cooling — the participants in the experimental group will receive a cold pack (gel pack, temperature -6 degrees to -12 degrees Celsius) will be placed on the target muscles for 20 minutes.
  Arms: Back cooling; Calf cooling; Hamstring cooling; Quadriceps cooling

SUMMARY:
This study aims to investigate the effects of localized muscle cooling on static and dynamic stability in healthy adults.

DETAILED DESCRIPTION:
Healthy young adult aged 18-30 years will be recruited from the College of Applied Medical Sciences (CAMS), King Saud University, Riyadh. Subjects will be excluded if they had a history of a hip or knee injury, sensory deficits in the lower extremity, a history of lower-extremity surgery, or a history of a quadriceps or hamstring muscle injury. The protocol was submitted to and approved by the Ethics Sub-Committee of Rehabilitation Research chair (RRC-2018-011). Participants will be requested to sign a written informed consent form approved by the institution ethics committee. A total of 50 participants were randomly assigned to the quadriceps cooling (QC: n = 10), hamstrings cooling (HC: n = 10), calf cooling (CC: n = 10), back muscle cooling (BC: n = 10) or control (no cooling: n = 10) group by a lottery method.A baseline assessment of mean center of gravity (COG), sway velocity (degrees/sec) for the unilateral Stance (US) will be performed. After the baseline assessment, a cold pack (gel pack, temperature -6 degrees to -12 degrees Celsius) will be placed on the target muscle for 20 minutes. One thin dry towel will be kept between the cold pack and the skin to prevent skin damage. Before and after the application of ice application the skin sensibility will be assessed by testing the participant's to a pinprick.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults

Exclusion Criteria:

* history of a hip or knee injury, sensory deficits in the lower extremity and lower back, a history of lower-extremity surgery, spinal surgery, or a history of a quadriceps or hamstring muscle injury.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
mean center of gravity (COG) sway velocity (degrees/sec) for the unilateral Stance (US) | up to 3 weeks
  The participants will be asked to stood in the marked position on the force plate, with their hands positioned on the iliac crests. The participants will be requested to lift the right foot to a standard height of 10 cm. This 10-second test will be performed three times in two test conditions, including eyes open (EO) and eyes closed (EC). The mean COG sway velocity (degrees/sec) from three trials of the US will be used in the analysis. The participants will be requested to perform the same test for the left leg. The US will be used to determine each participant's ability to maintain postural stability during unilateral standing in the EO and EC conditions.

CONTACTS AND LOCATIONS:
Overall Officials: AHMAD H ALGHADIR, PHD, Study Chair — King Saud University
Locations (1):
- RRC, KSU, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Data will be kept secure with the principal investigator (MR. SHAHNAWAZ ANWER) and sub-investigator (Dr. Ahmad Alghadir) due to confidentiality issues